CLINICAL TRIAL: NCT05746468
Title: The Mechanism and Effectiveness of Mindfulness-based Intervention for Reducing the Psychological Distress of Parents of Children With Autism Spectrum Disorder: An Ecological Momentary Intervention and Randomized Controlled Trial
Brief Title: Mindfulness Intervention for Parents of Children With ASD
Acronym: MAPASD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Xiaochen Zhou, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EC077/2223
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Mindfulness
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a combination of (1) a time-based system-triggered EMI, which will collect participants' sources and status of depression, anxiety and depression in daily life and provide instructions (audios and videos) on mindfulness practice, and (2) a longitudinal survey in parents of children with ASD. The participants will first complete a baseline questionnaire, and then participate in EMI via a smartphone application (App) for 8 consecutive weeks and receive the exercise prompts daily. The EMI will include questions of the self-reported feelings of depression, anxiety and depression. After the 8-week EMI, the participants will be invited to complete a post-experimental survey with similar questions in the baseline questionnaire. Two months after completing the EMI, participants will be contacted to complete a telephone follow-up survey with similar questions in the baseline questionnaire.
  Interventions: Behavioral: Ecological assessment and intervention
- Control group (Active Comparator): The control group will receive the longitudinal survey exactly the same as the intervention group and 8-week mindfulness-based short-messages sent by the research team on a daily basis. The messages will contain instructions of mindfulness-based practice which will be the same as the intervention group.
  Interventions: Behavioral: Audio-based Mindfulness intervention

INTERVENTIONS:
Behavioral: Ecological assessment and intervention — The MBI-EMI app will include five main parts, including virtual counselor, intervention library, weekly mindfulness practice, assessment bank and daily emotion log. In the eight weeks, the virtual counselor will initiate the conversation every day for three times (morning, afternoon and evening) to check the status of the participants. If the participants responded, the virtual counselor would invite the participants to rate their level of depression, stress and anxiety and then recommend appropriate mindfulness practice in the intervention library, such as 3-minute breathing space or mindful eating. The conversation between the virtual counselor and participants will be in the format of menu list and participants can easily choose from different options.
  Arms: Intervention group
Behavioral: Audio-based Mindfulness intervention — The control group will receive audio recordings of how to practice mindfulness at home.
  Arms: Control group

SUMMARY:
This study aims to develop a smartphone app based on mindfulness-based interventions and test its effectiveness in parents of children with ASD. This study aims:

1. To establish the relationship between different life events, cognitive appraisal, and the psychological distress between parents of children with autism spectrum disorder (ASD);
2. To demonstrate the relationship between parents' cognitive appraisal of life events and psychological distress moderated by mindfulness;
3. To examine the effectiveness of mindfulness-based intervention (MBI) via ecological momentary intervention (EMI) in reducing the psychological distress of parents of children with ASD;
4. To calculate the cost-effectiveness of MBI via EMI in reducing the psychological distress of parents of children with ASD.

DETAILED DESCRIPTION:
Existing studies have unequivocally demonstrated that parents of children with autism spectrum disorder (ASD) experience various daily life events and suffer from psychological distress. Mindfulness-based intervention (MBI) was found to be an effective buffer between parents' appraisal of life events and psychological distress. However, the mechanism behind the effectiveness was unclear, and traditional MBI in experimental settings were not tailored to personal real-life needs. This study proposed to conduct a randomized controlled trial (RCT) to examine the effectiveness and cost-effectiveness of MBI in the platform of ecological momentary intervention (EMI) in changing participants' cognitive appraisal of daily life events and reducing the psychological distress of parents of children with ASD.

This study aims to answer four research questions:

1. What's the relationship between participants' cognitive appraisal of their life events and psychological distress?
2. Will an increased level of mindfulness moderate the relationship between participants' cognitive appraisal of life events and psychological distress?
3. Will the participants who received MBI via EMI report significantly lower levels of psychological distress compared with those who did not?
4. Will the MBI via EMI be a more cost-effective option compared with the control group?

The proposed study will recruit 526 parents of children with ASD and randomly assign them into the intervention and control groups (263 in each group). Participants in the intervention group will install the EMI app on their smartphone. In the app, participants can browse different mindfulness exercises in the intervention bank at any time, talk to a virtual counselor and receive tailored mindfulness practice daily, practice formal mindfulness exercise every week, complete ecological momentary assessments on the cognitive appraisal of life events and receive a daily log of change of psychological status. Participants in the control group will only receive standardized mindfulness practice instructions 3 times/week. The effects of MBI will be assessed at the end of the intervention and at the 2-month follow-up.

The primary outcome will be participants' psychological distress measured by the depression anxiety stress scale. The secondary outcomes will include participants' subjective well-being, measured by the satisfaction with life scale, level of resilience measured by the psychological empowerment scale and the feasibility and acceptability of the EMI, measured by the treatment acceptability and adherence scale.

The potential benefit of the proposed study is to increase psychological well-being of parents of children with ASD and the method may extend to other participants in the future.

ELIGIBILITY:
The inclusion criteria will comprise

* parents of children with ASD (children aged between 6-18 and diagnosed with different functional levels of ASD by certified psychologists);
* own a mobile smartphone with internet access;
* will stay in Hong Kong during the 8-week EMI study period, and
* able to read and write in Chinese.

The exclusion criteria will include

* parents diagnosed with depression, anxiety, and stress disorder by certified doctors; and
* parents who do not live together with their children with ASD on the daily basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive Appraisal of Health Scale | right after the intervention
  The CAHS scale will be used to measure participants' cognitive appraisal of daily life events. This scale includes 28 items rated from 1 strongly disagree to 5 strongly agree. This scale was developed based on the transactional theory of stress and coping and thus consists of subscales of primary appraisal (threat, challenge, harm/loss and benign/irrelevant) and secondary appraisal. The internal consistency were all greater than .70.
Cognitive Appraisal of Health Scale | 2 months after the intervention
  The CAHS scale will be used to measure participants' cognitive appraisal of daily life events. This scale includes 28 items rated from 1 strongly disagree to 5 strongly agree. This scale was developed based on the transactional theory of stress and coping and thus consists of subscales of primary appraisal (threat, challenge, harm/loss and benign/irrelevant) and secondary appraisal. The internal consistency were all greater than .70.

SECONDARY OUTCOMES:
The Five Facet Mindfulness Questionnaire (FFMQ)-short version | right after the intervention
  will be used to measure participants' level of mindfulness before and after practicing. It includes 15 items measuring the five facets of mindfulness: observing, describing, acting with awareness, non-judging of inner experience and non-reactivity to inner experience. This scale was further validated and yield good convergent validity and internal consistency. The items will be rated using 1 (very rare)-5 (very often) Likert scale with higher score indicate higher level of mindfulness.
The Depression Anxiety Stress Scale | right after the intervention
  DASS is a self-report questionnaire that measures the emotional states of depression, anxiety, and stress. This scale contains 21 questions rated from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). There were seven questions for each one sub-scale of stress, depression, and anxiety. This scale showed good reliability (r=0.96 and 0.80 for the depression and anxiety subscales, respectively) and Cronbach's α was high for the three subscales in parents of children with ASD: 0.91 for the stress, 0.87 for anxiety, and 0.94 for depression and 0.92 for total scale. It has also been validated in Hong Kong population.
Satisfaction with Life Scale | right after the intervention
  The SWLS has 5 items scored on a 7-point scale (1 = strongly disagree to 7 = strongly agree) measuring participants' satisfaction with life and has a Cronbach's alpha for internal consistency of .87 and a test-retest correlation of .82. This scale has also been validated in Chinese and Hong Kong population.
Psychological Empowerment Scale for parents of children with a disability | right after the intervention
  It is a 32-item questionnaire on a 5-point scale (1 = strongly disagree to 5 = strongly agree) with four underlying sub-scales: (a) attitudes of control and competence, (b) cognitive appraisals of critical skills and knowledge, (c) formal participation in organizations, and (d) informal participation in social systems and relationships. This scale showed high reliability coefficients (.90-.97).

CONTACTS AND LOCATIONS:
Overall Officials: Qi Wang, Principal Investigator — Lingnan University

IPD SHARING:
Plan to Share IPD: Yes
The data of the primary and secondary outcomes will be shared
Supporting Information: Study Protocol
Time Frame: The data will be available after 6 months of the completion of the whole study.
Access Criteria: All scholars who can access the website.

REFERENCES:
- [Derived] Wang Q, Ng SM, Zhou X. The mechanism and effectiveness of mindfulness-based intervention for reducing the psychological distress of parents of children with autism spectrum disorder: A protocol of randomized control trial of ecological momentary intervention and assessment. PLoS One. 2023 Sep 13;18(9):e0291168. doi: 10.1371/journal.pone.0291168. eCollection 2023. PMID 37703248